CLINICAL TRIAL: NCT06178510
Title: POStoperative INTELLiVENT-adaptive Support VEntilation in Cardiac Surgery Patients II (POSITiVE II) - a Randomized Clinical Trial
Brief Title: I-ASV in Cardiac Surgery
Acronym: POSITiVE II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University Hospital Dubrava (Other); UniversitÃ degli Studi dell'Insubria (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Edda Tschernko, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: POSITiVE II v1.1
Record Dates: First submitted 2023-12-04; First posted 2023-12-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Ventilator Lung
Keywords: Adaptative Support Ventilation; INTELLiVENT; Cardiac Surgery; Workload

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTELLiVENT-ASV (Other): The ventilator set parameters such as tidal volume, respiratory rate, and positive end-expiratory pressure to ensure adequate ventilation and oxygenation. The investigators monitor it and define clinical target.
  Interventions: Device: INTELLiVENT-ASV.
- conventional ventilation (No Intervention): The investigators set and monitor parameters such as tidal volume, respiratory rate, and positive end-expiratory pressure to ensure adequate ventilation and oxygenation.

INTERVENTIONS:
Device: INTELLiVENT-ASV. — INTELLiVENT-ASV® is a closed-loop ventilation mode that automatically adjusts respiratory rate and tidal volume according to the oxygen and ventilatory patient needs
  Arms: INTELLiVENT-ASV

SUMMARY:
'POStoperative INTELLiVENT-adaptive support VEntilation in cardiac surgery patients II (POSITiVE II) is an investigator-initiated, international, multicenter, parallel, randomized clinical trial in patients after cardiac surgery.

DETAILED DESCRIPTION:
To compare INTELLiVENT-ASV with conventional ventilation with respect to (i.) quality of ventilation; and (ii.) ICU nursing staff workload in an international cohort of participants receiving postoperative ventilation after cardiac surgery. This study will also determine the effects of INTELLiVENT-ASV on clinical outcomes, including (iii.) duration of postoperative ventilation and (iv.) length of stay in ICU.

ELIGIBILITY:
Inclusion Criteria:

* 1. aged > 18 years of age;
* 2. scheduled for elective cardiac surgery; and
* 3. expected to receive postoperative ventilation in the ICU for > 2 hours.

Exclusion Criteria:

1. any emergency or semi-elective surgery (precluding informed written consent);
2. any surgery other than CABG, valve replacement or repair, or a combination (i.e., patients planned for surgery for congenital heart disease, or scheduled for heart transplantation are excluded);
3. enrolled in another interventional trail;
4. no written informed consent obtained;
5. history of recent pneumectomy or lobectomy;
6. history of COPD with oxygen at home;
7. body mass index > 35;
8. preoperative forced expiratory volume in the first second (FeV1)/forced vital capacity (VC) < 50% (if available);
9. preoperative arterial oxygen partial pressure (PaO2) < 60 mm Hg (at room air);
10. preoperative arterial carbon dioxide partial pressure (PaCO2) > 50 mm Hg;
11. preoperative left ventricular ejection fraction < 30% (if available);
12. preoperative systolic pulmonary artery pressure > 60 mm Hg (if available);
13. preoperative left ventricular mechanical support, e.g., Impella®; or
14. preoperative use of veno-venous or veno-arterial extracorporeal support

    At the end of surgery, patients are additionally excluded if a patient:
15. cannot be weaned from the extracorporeal support; or
16. unexpectedly needs implementation of an assist device

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of ventilation | During the first 2 hours, since admission on the ICU with the start of the intervention ventilation mode.
  The primary outcome is quality of ventilation, which is the proportion of time spent in three predefined and previously used zones of ventilation in the first 2 hours of postoperative ventilation.
  * An optimal zone = Tidal volume (TV) = 4-8 ml/kg of the predicted body weight (PBW) with an EtCO2 = 30-45mmHg, a plateau pressure = <31cmH2O and SpO2 = 93-98%.
  * An acceptable zone = TV = 8-12 ml/kg of PBW with an EtCO2 = 25-30 or 45-50mmHg, a plateau pressure = 31-35 cmH2O and SpO2 = 85-93% or >98%.
  * An unacceptable zone = TV >12 ml/kg of PBW or an EtCO2 = <25 or >50mmHg, plateau pressure >35 cmH2O or SpO2 = <85%.

SECONDARY OUTCOMES:
ICU nursing staff workload | 24 hours
  ICU nursing staff workload, which is captured by the ventilator software collecting data on alarms (number of alarms, types of alarm, duration of alarm, responses to alarm, alarm settings and adjustments, breath-by-breath alarm data, and any manual intervention at the ventilator) during postoperative care in the ICU
Duration of postoperative ventilation | 8 hours or until extubation
  The time from admission on the ICU until extubation.
Patient-ventilator asynchrony | Up to 6 hours of mechanical ventilation time
  patient-ventilator asynchrony requiring deepening of sedation and/or administration of muscle relaxants
Proportion of breath spent in zones of ventilation | Up to 6 hours of mechanical ventilation time
  Proportion of breaths spent in predefined and previously used zones of ventilation in the first 6 hours of postoperative ventilation.
  * An optimal zone = Tidal volume (TV) = 4-8 ml/kg of the predicted body weight (PBW) with an EtCO2 = 30-45mmHg, a plateau pressure = <31cmH2O and SpO2 = 93-98%.
  * An acceptable zone = TV = 8-12 ml/kg of PBW with an EtCO2 = 25-30 or 45-50mmHg, a plateau pressure = 31-35 cmH2O and SpO2 = 85-93% or >98%.
  * An unacceptable zone = TV >12 ml/kg of PBW or an EtCO2 = <25 or >50mmHg, plateau pressure >35 cmH2O or SpO2 = <85%.
ICU length of stay | From date of ICU admission until the date of ICU discharge, assessed up to 30 days
  Length of stay in the ICU
Hospital length of stay | From date of hospital admission until the date of hospital discharge, assessed up to 30 days
  Length of stay in hospital
Mortality | 28-day
  Mortality in ICU or hospital

CONTACTS AND LOCATIONS:
Overall Officials: Edda Tschernko, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
The results of the study will find their way into (inter-) national scientific journals and guidelines.
  We will submit a summary of results to scientific journals in the field of anesthesiology.

REFERENCES:
- [Derived] Bernardi MH, Bettex D, Buiteman-Kruizinga LA, de Bie A, Hoffmann M, de Kleijn J, Serafini SC, Molenaar MA, Paulus F, Persec J, Neto AS, Schuepbach R, Severgnini P, Sribar A, Schultz MJ, Tschernko E; POSITiVE II-investigators. POStoperative INTELLiVENT-adaptive support VEntilation in cardiac surgery patients (POSITiVE) II-study protocol of a randomized clinical trial. Trials. 2024 Jul 3;25(1):449. doi: 10.1186/s13063-024-08296-2. PMID 38961468